CLINICAL TRIAL: NCT02758912
Title: Open-label Clinical Pharmacokinetic Study of Cardionat®, Capsules 250 mg (JSC Nizhpharm, Russia) Using in Health Athlete Volunteers
Brief Title: Clinical Study of Medicinal Product Cardionat® Using in Health Athlete Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Burnasyan Federal Medical Biophysical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RU-FMBC-04-04-16
Record Dates: First submitted 2016-04-22; First posted 2016-05-03 (Estimated); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Stroke, Not Specified as Hemorrhage or Infarction; Angina Pectoris
MeSH Terms: conditions — Stroke; Angina Pectoris

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- arm 1, Cardionat® (Experimental): oral intake of study drug capsules at a dose of 1 g per day for 3 weeks.
  Interventions: Drug: оral intake of study drug capsules; study drug - Cardionat ® (trimethylhydrazinium propionate dihydrate), oral capsules 250 mg
- arm 2, Cardionat® (Experimental): oral intake of study drug capsules at a dose of 2 g per day for 3 weeks.
  Interventions: Drug: оral intake of study drug capsules; study drug - Cardionat ® (trimethylhydrazinium propionate dihydrate), oral capsules 250 mg

INTERVENTIONS:
Drug: оral intake of study drug capsules; study drug - Cardionat ® (trimethylhydrazinium propionate dihydrate), oral capsules 250 mg

SUMMARY:
The objective of this study is to evaluate the long-term plasma and urine pharmacokinetic parameters of Cardionat®, capsules 250 mg, when used in healthy athlete volunteers.

The study consists of four steps:

* Step 1. Screening - selecting healthy volunteers for inclusion in the study;
* Step 2. Assignment in one of the study group, prescription of the study drug;
* Step 3. Samples collections for pharmacokinetic analysis;
* Step 4. Evaluation of pharmacokinetic data.

DETAILED DESCRIPTION:
Cardionat is a structural analogue of gamma-butyrobetaine - a substance that is in every cell of the human body.

Under extra strain conditions cardionat restores the balance between oxygen delivery to the cell and cellular oxygen demand. Cardionat clears the intracellular accumulation of toxic metabolic products, protecting them from damage; also it has a general tonic effect. As a result of its use of the body acquires the ability to withstand stress and to quickly restore energy reserves. Because of these properties cardionat used to treat a variety of disorders of the cardiovascular system, disorders of blood supply to the brain, as well as to improve physical and mental performance. Synthesis of gamma-butyrobetaine, which has vasodilating properties, is highly increased as a result of reducing the concentration of carnitine.

In the case of acute ischemic myocardial injury cardionat slows the formation of necrotic areas, shortens the rehabilitation period.

In heart failure it increases myocardial contractility, increases exercise tolerance, reduces the frequency of angina attacks. In acute and chronic ischemic cerebrovascular disorders it improves blood circulation in the ischemic areas; it promotes blood redistribution increasing supply of the ischemic areas. It is effective in the case of vascular and dystrophic pathology of the ocular fundus. The drug eliminates functional disturbances of the nervous system in patients with chronic alcoholism during abstinence syndrome.

Pharmacokinetics After oral administration, the drug is rapidly absorbed. Bioavailability is 78%. The maximum plasma concentration is reached 1-2 hours after oral ingestion. The drug is metabolized in the body with the formation of two major metabolites, which are excreted by the kidneys. The half-life after oral intake is dose-dependent, and is usually 3 to 6 hours.

Indications for use:

As a part of combination treatment of coronary heart disease (angina, myocardial infarction), congestive heart failure and dyshormonal cardiomyopathy, as well as part of combination treatment of acute and chronic cerebrovascular disorders (stroke and cerebrovascular insufficiency).

Reduced working capacity; physical stress, including physical stress in athletes.

Abstinence syndrome in chronic alcohol abusers (in combination with specific alcohol abuse therapy).

In this study, volunteers will receive study medication in the form of oral capsules 250 mg.

The study drug will be applied as follows:

* Group 1: intake of study medication capsules orally at a dose of 1 g per day for 3 weeks - 14 volunteers (7 males and 7 females);
* Group 2: intake of study medication capsules at a dose of 2 g per day for 3 weeks - 14 volunteers (7 males and 7 females).

Study results will be published in "Drug Testing and Analysis" journal

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers of both sexes aged 18 to 35 years old, caucasians;
2. At least 1st sports category among adults;
3. Verified diagnosis "healthy" according to a detailed medical history, and according to standard clinical, laboratory and instrumental methods of examination;
4. BMI should be between 18.5 to 30 kg / m2;
5. Signed Volunteer information sheet with the Informed consent form;
6. Agreement of volunteer to use adequate methods of contraception (contraceptive reliability over 90%: the cervical cap with spermicide, diaphragm with spermicide, condoms, intrauterine devices), or total abstinence from sexual activity for the period of the study:

   * For women during the whole period from 30 days prior to the signing a Volunteer's information sheet with Informed consent form to 30 days after completion of study participation; in the period from the date of signing the Informed consent up to 30 days after completion of study participation barrier method of contraception should be used, if it is not the main method;
   * For men during the whole period from signing a Volunteer's information sheet with the Informed consent form and until the completion of the study barrier method of contraception should be used.

Non - inclusion criteria:

1. Allergy in the past;
2. Drug intolerance, hypersensitivity to any component of the study drug;
3. Chronic cardiovascular, bronchopulmonary, endocrine or nervous systems diseases (including psychiatric disorders), and diseases of the gastrointestinal tract (GIT), liver, kidney, blood disorders, surgical interventions on the gastrointestinal tract (except appendectomy);
4. Fructose intolerance, glucose-galactose malabsorption or sucrase-isomaltase insufficiency;
5. Poor developed superficial veins of the forearm;
6. Acute infectious, non-infectious and allergic diseases in less than 4 weeks prior to Visit 1 (screening);
7. Positive blood test for HIV, syphilis, hepatitis B and C;
8. Intake of more than 10 units of alcohol per week (1 unit of alcohol is equivalent to 1/2 liters of beer, 200 ml wine or 50 ml of spiritus) alcoholism, drug addiction or drug abuse in the past;
9. Smoking more than 10 cigarettes per day;
10. Systolic blood pressure measured in the "sitting" position below 100 mm Hg or above 130 mm Hg and/or diastolic blood pressure below 60 mm Hg or above 90 mm Hg;
11. Heart rate below 40 beats / min;
12. Any deviation from the normal range of the results of clinical and laboratory tests (complete blood count, urinalysis, blood chemistry) and instrumental tests (ECG);
13. Intake of any medicines, including any supplements, not agreed with study doctor;
14. Blood donation: 0-49 ml - 0 days prior to Visit 1 (screening); 50-449 ml - in less than 30 days prior to Visit 1; 450-800 ml or more - less than 60 days prior to Visit 1; 800 ml - by the decision of the Chief Investigator, if the period of time prior to the visit 1 is more than 60 days;
15. Plasmapheresis in less than 14 days prior to Visit 1;
16. Participation in the competitions, where doping tests are required, while participating in this clinical trial (within 6 ± 2 months from the date of inclusion in the study - Visit 1 (Screening));
17. Participation in the study of another medicinal product or medical device in less than 3 months prior to the study;
18. Volunteer's inability or unwillingness to comply with the study protocol requirements;
19. Any reason, which, according to researcher opinion, will impede the participation of volunteer in the study;
20. Pregnant or lactating women (all women should have a negative pregnancy test results on the day of screening).

Exclusion Criteria:

1. Unexpected and previously unknown adverse reactions (if it is related to support volunteer's health);
2. Occurrence of SAEs;
3. Acute diseases or conditions that are not SAEs, but according to researchers opinion, require exclusion of volunteers from the study;
4. Decision to volunteer to withdraw from the study;
5. Violation by volunteer of prescribed regimen and violation of research restrictions (by the decision of the investigator);
6. Investigator's decision to exclude the volunteer from the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-11; Primary Completion 2019-09-25 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 3 weeks after assignment of all eligible volunteers to one of the study groups (day 22th)
  Data collected and assessed for each AE include type, duration, relationship to study drug, action taken and the outcome of the event. Registration of SAEs begins right after the first dose of study drug during the whole course of treatment.

SECONDARY OUTCOMES:
Cardionat® levels in blood | following days 0, 22, 26, 33, 40(twice), 41, 47(twice), 48, 54(twice), 55, 61(twice), 62, 75(twice), 76, 89(twice), 90, 103(twice), 104, 133(twcie), 134, 150(twice), 151
  Test drug (Cardionat®) concentration in blood plasma of healthy volunteers after its oral administration during a period of 21 days (3 weeks) at doses of 1000 mg and 2000 mg (Group 1 and 2, respectively) by a validated HPLC method.
Cardionat® levels in urine | following days 0, 22, 26, 33, 40(twice), 41, 47(twice), 48, 54(twice), 55, 61(twice), 62, 75(twice), 76, 89(twice), 90, 103(twice), 104, 133(twcie), 134, 150(twice), 151
  Test drug (Cardionat®) concentration in urine of healthy volunteers after its oral administration during a period of 21 days (3 weeks) at doses of 1000 mg and 2000 mg (Group 1 and 2, respectively) by a LC/MS/MS method using a liquid chromatograph Eksigent ekspert ultraLC 100 and a tandem mass spectrometer AB Sciex QTrap 3200.
Exercise load duration (Tel) | following days 22, 26, 33, 40, 41, 47, 48, 54, 55, 61, 62, 75, 76, 89, 90, 103, 104, 133, 134, 150, 151
  Exercise load duration (tel) is determined from the beginning of the test until termination by the athlete after the appearance of subjective impossibility to continue to carry the load - testing "to failure."
Time of onset of aerobic threshold (Tat) | following days 22, 26, 33, 40, 41, 47, 48, 54, 55, 61, 62, 75, 76, 89, 90, 103, 104, 133, 134, 150, 151
  Time of onset of aerobic threshold (tat) is a time-point of exercise load test where energy supplied primarily by aerobic glycolysis. It corresponds to a level of homeostasis, in which an increase in lactate occurs in the blood, exceeding a certain baseline level (up to this point lactate appearing in the muscles was completely neutralized by buffer systems). It is determined during the test at a value of the respiratory quotient of R ~ 0,85, corresponding to the appearance of the first bend on oxygen consumption-time curve (pulmonary ventilation).
Time of onset of the anaerobic threshold (Tant) | following days 22, 26, 33, 40, 41, 47, 48, 54, 55, 61, 62, 75, 76, 89, 90, 103, 104, 133, 134, 150, 151
  Time of onset of the anaerobic threshold (tant) is a time-point of exercise load test where anaerobic glycolysis becomes the leading mechanism of energy supply, and persistent accumulation of lactate with increase of lactate / pyruvate ration in muscle and arterial blood are observed. It is determined during the test at a value of the respiratory quotient of R ~ 1,01, corresponding to the appearance of the second bend on oxygen consumption-time curve (pulmonary ventilation).
Respiratory quotient (R) | following days 22, 26, 33, 40, 41, 47, 48, 54, 55, 61, 62, 75, 76, 89, 90, 103, 104, 133, 134, 150, 151
  Respiratory quotient (R) is a ratio of carbon dioxide volume emitted from the body to the volume of the absorbed oxygen during that time. Respiratory quotient is increased during intensive work load effort and lung hyperventilation, when additional previously binded CO2 is released from the body.
Maximum oxygen consumption (MOC) | following days 22, 26, 33, 40, 41, 47, 48, 54, 55, 61, 62, 75, 76, 89, 90, 103, 104, 133, 134, 150, 151
  The absolute criterion of achieving the level of maximum oxygen consumption is the presence of a "plateau" on a curve of oxygen consumption from the load power dependence. Indirect criteria of achieving the MOC include: a significant increase of lactate; Respiratory quotient ≥1,11 increase of heart rate to 180-200 beats/min.
The level of oxygen consumption in the aerobic threshold (V'O2AT) | following days 22, 26, 33, 40, 41, 47, 48, 54, 55, 61, 62, 75, 76, 89, 90, 103, 104, 133, 134, 150, 151
  The level of oxygen consumption in the aerobic threshold, AT (V'O2AT) is determined at the time of the onset of aerobic threshold
The level of oxygen consumption in the anaerobic threshold (V'O2ANT) | following days 22, 26, 33, 40, 41, 47, 48, 54, 55, 61, 62, 75, 76, 89, 90, 103, 104, 133, 134, 150, 151
  The level of oxygen consumption in the anaerobic threshold, ANT (V'O2ANT) is determined at the time of the onset of anaerobic threshold
Heart rate (HR) | following days 22, 26, 33, 40, 41, 47, 48, 54, 55, 61, 62, 75, 76, 89, 90, 103, 104, 133, 134, 150, 151
  Heart rate (HR) is registered during the whole testing period (HRres, HRat, HR ANT, HR max, HR recovery), which allows to get the pulse profile, not only for a particular athlete, but also for the contingent of the same sports and qualification level.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Budget Institution "State Scientific Center of Russian Federation - the Federal Medical Biophysical Center named after A I Burnazyan" (FSBI SSC FMBC name AI Burnazyan FMBA of Russia), Moscow, Russia

REFERENCES:
- [Background] Rabin O, Uiba V, Miroshnikova Y, Zabelin M, Samoylov A, Karkischenko V, Semyonov S, Astrelina T, Razinkin S. Meldonium long-term excretion period and pharmacokinetics in blood and urine of healthy athlete volunteers. Drug Test Anal. 2019 Apr;11(4):554-566. doi: 10.1002/dta.2521. Epub 2018 Nov 12. PMID 30328291